CLINICAL TRIAL: NCT06642649
Title: Evaluation and Comparison Between General Anesthesia VS Two Types of Combined Anesthesia (general and Spinal Anesthesia) for Opioid Consumption in Laparoscopic Hysterectomy: a Multi-Center, Randomized, Prospective, Controlled Trial
Brief Title: Evaluation and Comparison Between General Anesthesia VS Two Types of Combined Anesthesia for Opioid Consumption in Laparoscopic Hysterectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Andrea Saporito (Other)
Responsible Party: Sponsor-Investigator, Andrea Saporito, Head of Anesthesiology, Prof.Dr.Med., Ente Ospedaliero Cantonale, Bellinzona
Organization: Ente Ospedaliero Cantonale, Bellinzona (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LpsSa
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2024-10

CONDITIONS: Laparoscopic Hysterectomy; Gynecology
Keywords: laparoscopic hysterectomy; spinal anesthesia; general anesthesia
MeSH Terms: interventions — Anesthesia, General; Control Groups; Anesthetics, Local; Fentanyl

STUDY DESIGN:
Intervention Model Description: randomized, controlled, prospective, multi-center
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- study intervention with spinal anesthesia composed by local anesthetic, morphine and no fentanyl (Active Comparator): Every patient will receive, before induction of general anesthesia as in control group, a spinal anesthesia composed by hyperbaric bupivacaine 5 mg 0,5% and morphine sulfate 100 mcg.
  Interventions: Procedure: General Anesthesia + Spinal anesthesia combined (local anesthetic, morfine and no fentanyl)
- study intervention with spinal anesthesia composed by local anesthetic, morphine and 20 mcg fentanyl (Active Comparator): every patient will receive, before induction of general anesthesia, as in the control group, a spinal anesthesia composed by hyperbaric bupivacaine 5 mg 0,5%, morphine sulfate 100 mcg and fentanyl 20 mcg.
  Interventions: Procedure: General Anesthesia + Spinal anesthesia combined (local anesthetic, morfine and 20 mcg fentanyl)
- study intervention NO spinal (Active Comparator): Every patient will receive a general anesthesia induced with propofol (1.5-2.5 mg/kg, individually adjusted), rocuronium (0.6 mg/kg) for muscle relaxation and a continuous infusion of remifentanil (0.05-0.3 mcg/kg/min, depending on the clinical characteristics of the patient). General anesthesia was maintained with a continuous infusion of propofol (4-8 mg/kg/h), and the infusion of remifentanil which was started with the induction. Fractionated doses of rocuronium were administered based on TOF monitoring (train of four) to maintain muscle relaxation.
  Interventions: Procedure: General Anesthesia (control group)

INTERVENTIONS:
Procedure: General Anesthesia (control group) — Only General Anestesia
  Arms: study intervention NO spinal
Procedure: General Anesthesia + Spinal anesthesia combined (local anesthetic, morfine and no fentanyl) — General anesthesia + spinal anesthesia with local anesthetic and morfine
  Arms: study intervention with spinal anesthesia composed by local anesthetic, morphine and no fentanyl
Procedure: General Anesthesia + Spinal anesthesia combined (local anesthetic, morfine and 20 mcg fentanyl) — General anesthesia + spinal anesthesia with local anesthetic, morfine and fentanyl
  Arms: study intervention with spinal anesthesia composed by local anesthetic, morphine and 20 mcg fentanyl

SUMMARY:
The aim of the study is to evaluate and compare general anesthesia VS two types of combined anesthesia in opioid consumption after laparoscopic hysterectomy

DETAILED DESCRIPTION:
Managing post-operative pain is essential to reduce length of stay, complications, mortality, healthcare costs and the risk of readmission to hospital. At the same time, pain treatment, especially with opiod drugs, could cause side effects and worsen the quality of post-operative hospitalization. Furthermore, intrathecal fentanyl may cause an acute tolerance to opioids, and may worsen postoperative analgesia. In literature, some studies underline how the use of regional anesthesia represents an effective solution in pain control. The goal of this study would be to determine whether post-operative analgesic needs and pain levels are increased by mixing intrathecal fentanyl with spinal anesthesia and intrathecal morphine.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 year of age,
* ASA physical status I to III scheduled for laparoscopic hysterectomy (with or without adnexectomy)

Exclusion Criteria:

* patients with inability to consent,
* patient refusal,
* contraindication to spinal anesthesia (e.g., hemodynamic instability, infection at the surgery site, and neurologic defects such as transverse myelitis, coagulopathies or ongoing anticoagulant therapy),
* known chronic pain syndrome, known
* suspected non- compliance,
* drug, or alcohol abuse ,
* major oncological surgeries,
* allergy to drugs used in the protocol,
* previous chronic use of analgesics
* history of opioid abuse

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 45 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
PCA morphine consumption in the first 24 and 48 postoperative hours | 48 hours

SECONDARY OUTCOMES:
Number of patients with intraoperative hypotension (MAP e amine) | during surgery
intraoperative opioids consumption | during surgery
postoperative pain scores (VAS) - Visual Analogue Scale - at 4, 12, 24 and 48 hours (from 0 to 10) | 48 hours
postoperative pruritus (rating 1-10) | 48 hours
Number of patientes with postoperative nausea and vomiting | 48 hours
  At the time of the visit, the patient will be asked if any episodes of nausea or vomiting have occurred (in the concept of a dichotomous variable YES or NO) and if these have required the administration of antiemetic drugs. The number of episodes and the number of requests for drugs in reserve for management will be reported
Number of patients with urinary retention | 48 hours
  At the time of the visit, once the bladder catheter has been removed after the operation, the patient and the care staff will be asked if any episodes of urinary retention have occurred (in the concept of a dichotomous variable YES or NO) and if further treatment has been necessary. bladder catheterization.
Quality of Recovery (QoR-15 Score) (0 to 150) | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Saporito, Anesth, Study Chair — Ente Ospedaliero Cantonale, Bellinzona
Locations (2):
- Switzerland (2):
  - Ente Ospedaliero Cantonale ORBV, Bellinzona, Switzerland
  - Ente Ospedaliero Cantonale, Ospedale Regionale di Bellinzona e Valli, Bellinzona, Switzerland

IPD SHARING:
Plan to Share IPD: No